CLINICAL TRIAL: NCT04451473
Title: The Short Term and Long Term Comparison of Lung Surgery With or Without Enhanced Recovery
Brief Title: Lung Surgery With Enhanced Recovery VS. Lung Surgery Without Enhanced Recovery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ERAS ZYP
Record Dates: First submitted 2020-06-27; First posted 2020-06-30 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-02

CONDITIONS: Lung Cancer; Surgery; ERAS
MeSH Terms: conditions — Lung Neoplasms | interventions — Enhanced Recovery After Surgery

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS- Group (Experimental): Patients underwent surgery for lung cancer accepted the enhanced recovery after surgery (ERAS).
  Interventions: Procedure: Enhanced Recovery After Surgery (ERAS )
- Control- Group (Other): Patients underwent surgery for lung cancer without enhanced recovery after surgery (ERAS).
  Interventions: Procedure: Traditional perioperative management without Enhanced Recovery After Surgery (ERAS )

INTERVENTIONS:
Procedure: Enhanced Recovery After Surgery (ERAS ) — the treatment of procedure according to Guidelines for enhanced recovery after lung surgery: recommendations of the ERAS Society and the ESTS
  Arms: ERAS- Group
Procedure: Traditional perioperative management without Enhanced Recovery After Surgery (ERAS ) — the treatment of procedure not abiding Guidelines for enhanced recovery after lung surgery
  Arms: Control- Group

SUMMARY:
Objective: The adoption of Enhanced Recovery Surgery programs in lung resection is relatively recent with limited outcome data. This study aimed to determine the impact of an Enhanced Recovery Surgery pathway on short- term and long- term results in patients undergoing lung resection for primary lung cancer.

Methods: A Randomized Controlled Trial was designed to collect the perioperative data on consecutive patients undergoing lung resection for primary lung cancer. Patients will be randomizely assigned to the ERAS- Group and Control- Group. Short-term and long- term effect will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria: patients with stage I-IIIa Non-small-cell Lung Cancer underwent radical resection or other benign lung lesions need VATS surgery.

-

Exclusion Criteria: cardio-pulmonary function couldn't tolerate surgery

-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2019-10-08 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
intensive care unit utilization | within 4 days after surgery
  the time in intensive care unit utilization
the degree of pain | within 4 days after surgery
  Visual Analogue Scale/Score
the time of ambulation | within 48 hours after surgery
  the time after surgery that patients could leave the bed and walk
the time for oral feed | within 48 hours after surgery
  the time for oral feed
the time of hospitalization | within 5 days after surgery
  the time of hospitalization
complications | within 7 days after surgery
  the rate of complications

SECONDARY OUTCOMES:
disease- free survival | within 5 years after surgery
  disease- free survival
overall survival | within 10 years after surgery
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Xiaogang Zhao, Doctor, Study Director — The Second Hospital of Shandong University
Locations (1):
- Yunpeng Zhao, Jinan, Shandong, China

REFERENCES:
- [Derived] Ding Y, Zhou L, Shan L, Zhang W, Li P, Cong B, Tian Z, Zhao Y, Zhao X. Video- assisted thoracoscopic lung resection with or without enhanced recovery after surgery: a single institution, prospective randomized controlled study. Front Oncol. 2024 Nov 8;14:1474438. doi: 10.3389/fonc.2024.1474438. eCollection 2024. PMID 39582544